CLINICAL TRIAL: NCT06930157
Title: Multi-center Randomized Controlled Clinical Study of Shenling Baishu Granule to Prevent the Recurrence of Low-risk Colorectal Adenoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Affiliated Hospital of Nanjing University of Chinese Medicine (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Sixth Affiliated Hospital, Sun Yat-sen University (Other); Shuguang Hospital of Shanghai University of Traditional Chinese Medicine (Unknown); Beijing Friendship Hospital (Other); Yueyang Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Institute of Science, Beijing Tongrentang Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Xiaobo Li, Principal Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KY2024-191-C
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Low-risk Colorectal Adenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Shenling Baizhu Granules) (Experimental): Participants will take Shenling Baizhu granules (6 g, three times daily) for 6 months, started within 3 months after standard endoscopic treatment, in addition to basic health education.
  Interventions: Drug: Shenling Baizhu granules (TCM patent medicine)
- Control Group (No intervention) (No Intervention): Participants will receive only basic health education without taking Shenling Baizhu granules.

INTERVENTIONS:
Drug: Shenling Baizhu granules (TCM patent medicine) — Shenling Baizhu granules is a traditional Chinese medicine preparation in granular form. Participants in the experimental group will take 6 g orally three times daily for 6 months, initiated within 3 months after baseline endoscopic resection and health education. The granules should be taken before meals or at the same time as eating. The granules contain multiple Chinese herbs including Ginseng, Poria, Atractylodes macrocephala, and other traditional ingredients. This formulation is standardized according to Chinese pharmacopoeia standards and is manufactured under GMP conditions. This intervention is being tested for its ability to prevent the recurrence of low-risk colorectal adenomas after endoscopic resection.
  Arms: Experimental Group (Shenling Baizhu Granules)

SUMMARY:
1. Complete a large-sample, multicenter, randomized blank-controlled clinical trial to evaluate Shenling Baizhu Granules for the prevention of colorectal adenoma recurrence.
2. Generate high-level, internationally recognized clinical evidence to support the development of clinical practice guidelines for the prevention and treatment of colorectal adenoma using traditional Chinese medicine, and to strengthen the recommendation level of Shenling Baizhu Granules in clinical guidelines.
3. Define the clinical characteristics of patient subgroups most likely to benefit from Shenling Baizhu Granules for preventing colorectal adenoma recurrence.

DETAILED DESCRIPTION:
This study is designed within the traditional Chinese medicine (TCM) framework for colorectal adenoma and will be conducted as a prospective, multicenter, open-label, randomized, blank-controlled clinical trial. All participants will undergo standard endoscopic minimally invasive treatment and receive health education. In addition to these measures, participants in the intervention group will receive Shenling Baizhu Granules (6 g per dose, three times daily). The intervention will be initiated within 3 months after the baseline treatment/health education and continued for 6 consecutive months. Participants in the control group will not receive Shenling Baizhu Granules.

At baseline, demographic characteristics, adenoma-related information, and TCM syndrome assessment scores will be collected. Follow-up will be conducted every 6 months during the first 2 years, and once in the third year. Biospecimens and TCM assessments will be collected at three time points: (i) baseline, (ii) 6 months after initiation of medication in Year 1, and (iii) after colonoscopic reassessment in Year 3. At each time point, plasma, stool, tongue coating, saliva, and tissue samples, as well as the TCM syndrome assessment questionnaire, will be obtained.

To characterize the subpopulation most likely to benefit from Shenling Baizhu Granules in preventing colorectal adenoma recurrence, we will integrate and analyze: baseline clinical factors (e.g., age, sex, family history of cancer, smoking and alcohol use); conventional medical features (e.g., adenoma location, number, size, histopathological type, and concomitant medications); TCM-related features (e.g., evolution of TCM syndrome patterns and objective tongue/pulse parameters); and biological profiles (e.g., cytokines, proteins, metabolites, and gut microbiota). Common characteristics of the beneficial population will then be summarized based on these multidimensional data.

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for low-risk colorectal adenoma.
* Has undergone a colonoscopy of adequate quality (adequate bowel preparation, cecal intubation achieved, and withdrawal time ≥6 minutes) and received endoscopic minimally invasive polypectomy.
* Within 3 months after adenoma resection.
* 18-70 years of age; any sex.
* Willing to participate and has voluntarily provided written informed consent.

Exclusion Criteria:

* Incomplete adenoma resection.
* Long-term use of aspirin, folic acid, calcium supplements, vitamin D, or similar agents.
* Known hereditary polyposis syndromes (e.g., familial adenomatous polyposis) or hereditary colorectal cancer syndromes (e.g., Lynch syndrome/hereditary nonpolyposis colorectal cancer).
* Colonoscopy findings strongly suggestive of inflammatory bowel disease.
* History of malignancy within the past 5 years.
* Pregnant or breastfeeding women, or participants with pregnancy potential who are planning pregnancy.
* Severe cardiovascular or cerebrovascular disease, hepatic or renal insufficiency, or diabetes mellitus.
* Severe psychiatric disorders that would preclude cooperation with colonoscopy procedures.
* Current condition preventing oral administration of the study drug (e.g., dysphagia, chronic diarrhea, intestinal obstruction).
* Participation in another clinical study within the past 3 months or current participation in another clinical study.
* Any other condition that, in the investigator's judgment, makes the participant unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of metachronous low-risk adenomas within 3 years after first dose | At 3 years after enrollment
  The incidence of metachronous low-risk adenomas will be calculated for each group as the number of participants with metachronous low-risk adenomas detected on surveillance colonoscopy within 3 years of enrollment divided by the total number of participants in that group.

SECONDARY OUTCOMES:
Colorectal adenoma progression rate | At 3 years after enrollment
  The progression rate will be calculated for each group as the number of participants in whom colorectal adenoma progression (defined as high-risk adenoma and/or malignant transformation) is detected on surveillance colonoscopy within 3 years after enrollment divided by the total number of participants in that group.
TCM syndrome score | At baseline, 6 months, and 36 months
  The Traditional Chinese Medicine Syndrome Survey assesses bowel habits, abdominal symptoms, and secondary symptoms like oral discomfort and appetite, with scores ranging from 0 (no symptoms) to higher values indicating increasing severity, alongside tongue and pulse observations.

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No